CLINICAL TRIAL: NCT04149405
Title: Investigation of the Effects of Bisphosphonate on the Gingival Crevicular Fluid Levels of Sclerostin and the DKK-1 in Individuals With Postmenopausal Osteoporosis With Periodontal Changes
Brief Title: Alterations of GCF Levels of Sclerostin and DKK-1 in Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Feyza Otan ÖZDEN, Principal Investigator, Ondokuz Mayıs University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KAEK 2016/100
Record Dates: First submitted 2019-10-12; First posted 2019-11-04 (Actual); Results first posted 2020-12-01 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2020-11

CONDITIONS: Osteoporosis, Postmenopausal; Periodontitis
Keywords: sclerostin; dickkopf-related protein-1
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Periodontitis; Sclerosteosis | interventions — Periodontal Index

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group A (Active Comparator): * Subjects with chronic periodontitis and osteoporosis.
  * Phase 1 periodontal therapy and bisphosphonate therapy ( Aclasta: intravenous infusion of 5 mg of zoledronic acid once a year) were administered to the subjects.
  Interventions: Procedure: Phase 1 periodontal therapy; Drug: Bisphosphonate therapy
- Group B (Active Comparator): * Subjects with chronic periodontitis and systemically healthy.
  * Phase 1 periodontal theraphy was administered to the subjects.
  Interventions: Procedure: Phase 1 periodontal therapy
- Group C (Active Comparator): * Subjects with periodontally healthy and osteoporosis.
  * Bisphosphonate therapy ( Aclasta: intravenous infusion of 5 mg of zoledronic acid once a year) were administered to the subjects.
  Interventions: Drug: Bisphosphonate therapy
- Group D (No Intervention): * Systemically and periodontally healthy controls
  * No intervention has been made.

INTERVENTIONS:
Procedure: Phase 1 periodontal therapy — Scaling and root planning with ultrasonic and hand instruments under local anesthesia.
  Other Names: Periodontal treatment
  Arms: Group A; Group B
Drug: Bisphosphonate therapy — Using aclasta: intravenous infusion of 5 mg of zoledronic acid once a year
  Other Names: Osteoporosis treatment
  Arms: Group A; Group C

SUMMARY:
Symptoms of periodontal disease are tissue destruction and destruction of the alveolar bone which supports the tooth. Wnt way (wingless-type MMTV integration site family) plays a role in the regulation of bone homeostasis in periodontal disease-induced bone resorption. The Wnt / β-catenin signal is controlled by physiological antagonists, including dickkopf released from osteocytes-associated protein 1 (DKK-1) and sclerostin (SOST). Thus, Wnt inhibitors SOST and DKK-1 affect bone mass changes. Bisphosphonates used in osteoporous treatment are selective inhibitors of bone resorption. In the serum of postmenopausal osteoporotic women treated with bisphosphonate, short-term and decreased DKK-1 level during the treatment, and increased SOST in the late period were reported. Increased bone formation after bisphosphonate treatment in postmenopausal osteoporotic patients has been associated with increased serum SOST level. The aim of our study is to investigate the effect of bisphosphonate in patients with post-menopausal osteoporosis on the bone demolition metabolism in periodontally healthy and periodontally diseased tooth regions and gingival health with the clinical data by investigating the SOST and DDK-1 molecules that play role in bone destruction mechanism.

DETAILED DESCRIPTION:
This study aims to reveal the effect of initial periodontal treatment together with bisphosphonate on sclerostin (SOST) and dickkopf-related protein-1 (DKK-1) in gingival crevicular fluid (GCF) of patients with osteoporosis.

Clinical recordings and GCF were obtained from postmenopausal women; with chronic periodontitis and those using bisphosphonate (Group A, n=12), with chronic periodontitis and otherwise healthy (Group B, n=10), without chronic periodontitis and those using bisphosphonate (Group C, n=11), systemically and periodontally healthy controls (Group D, n=10) at the baseline.

GCF sampling were recorded and repeated at the 6th and 12th months in Group A, B and C. SOST and DKK-1 values were measured by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Women with T scores less than -2.5 (groups A and C)
* The periodontitis patients were selected based on the radiographical evidence of bone loss, presence of four or more sites with bleeding on probing (BOP), ≥5 mm pocket depth (PD) and ≥6 mm clinical attachment loss (CAL).
* The clinically healthy control groups were selected on the basis of no radiographic bone loss or CAL and PD≤3 mm.

Exclusion Criteria:

* Any known systemic disease rather than osteoporosis
* Smoking
* Antibiotic therapy within the last 3 months
* Periodontal treatment in the last 6 months

Ages: 51 Years to 66 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2018-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eser Acarel, PhD,Prof.Dr., Study Director — Ondokuz Mayıs University, School of Dentistry, Department of Periodontology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hampson G, Edwards S, Conroy S, Blake GM, Fogelman I, Frost ML. The relationship between inhibitors of the Wnt signalling pathway (Dickkopf-1(DKK1) and sclerostin), bone mineral density, vascular calcification and arterial stiffness in post-menopausal women. Bone. 2013 Sep;56(1):42-7. doi: 10.1016/j.bone.2013.05.010. Epub 2013 May 20. PMID 23702386
- [Background] Papapoulos SE, Landman JO, Bijvoet OL, Lowik CW, Valkema R, Pauwels EK, Vermeij P. The use of bisphosphonates in the treatment of osteoporosis. Bone. 1992;13 Suppl 1:S41-9. doi: 10.1016/s8756-3282(09)80009-4. PMID 1581119
- [Background] Juluri R, Prashanth E, Gopalakrishnan D, Kathariya R, Devanoorkar A, Viswanathan V, Romanos GE. Association of Postmenopausal Osteoporosis and Periodontal Disease: A Double-Blind Case-Control Study. J Int Oral Health. 2015 Sep;7(9):119-23. PMID 26435630
- [Result] Lane N, Armitage GC, Loomer P, Hsieh S, Majumdar S, Wang HY, Jeffcoat M, Munoz T. Bisphosphonate therapy improves the outcome of conventional periodontal treatment: results of a 12-month, randomized, placebo-controlled study. J Periodontol. 2005 Jul;76(7):1113-22. doi: 10.1902/jop.2005.76.7.1113. PMID 16018754
- [Result] Balli U, Aydogdu A, Dede FO, Turer CC, Guven B. Gingival Crevicular Fluid Levels of Sclerostin, Osteoprotegerin, and Receptor Activator of Nuclear Factor-kappaB Ligand in Periodontitis. J Periodontol. 2015 Dec;86(12):1396-404. doi: 10.1902/jop.2015.150270. Epub 2015 Sep 14. PMID 26367496
- [Result] Napimoga MH, Nametala C, da Silva FL, Miranda TS, Bossonaro JP, Demasi AP, Duarte PM. Involvement of the Wnt-beta-catenin signalling antagonists, sclerostin and dickkopf-related protein 1, in chronic periodontitis. J Clin Periodontol. 2014 Jun;41(6):550-7. doi: 10.1111/jcpe.12245. PMID 24576302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal women who were admitted to Ondokuz Mayıs University (OMU), Faculty of Medicine, Department of Endocrinology and Metabolism between 2016 and 2018.
  Patients eligible for the study were directed to OMU, Faculty of Dentistry, Department of Periodontology for periodontal examination after obtaining medical records.
Pre-assignment Details: Smokers and subjects who had received antibiotic treatment in the last 3 months and/or periodontal treatment in the last 6 months were excluded from the study.
Groups:
- Group A: subjects with chronic periodontitis and osteoporosis
- Group B: subjects with chronic periodontitis and systemically healthy
- Group C: subjects with periodontally healthy and osteoporosis
- Group D: systemically and periodontally healthy controls
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D
Started | 12 | 10 | 11 | 10
Completed | 12 | 10 | 11 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Total
Number analyzed (Participants) | 12 | 10 | 11 | 10 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.67 (4.77) | 57.00 (4.39) | 56.45 (3.88) | 56.30 (3.91) | 56.88 (4.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 11 | 10 | 43
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 12 | 10 | 11 | 10 | 43
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 12 | 10 | 11 | 10 | 43
baseline sost values [Mean (Standard Deviation); unit: ng/ml] — initial sclerostin values
  ng/ml | 494.096 (99.840) | 634.731 (152.554) | 1023.071 (512.733) | 2131.87 (485.784) | 1103.417 (751.080)
baseline dkk-1 levels [Mean (Standard Deviation); unit: ng/ml] — initial dickkopf-related protein-1 values
  ng/ml | 1031.323 (506.985) | 1264.632 (492.691) | 2630.430 (1679.080) | 4269.394 (1734.732) | 2358.505 (1801.692)

OUTCOME MEASURES:

1. Primary Outcome: Sost Values for 6th Month
Description: levels of sclerostin in 6th month
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Group A: scaling and root planning, bisphosphonate therapy (zoledronic acid)
  periodontal phase 1 therapy: periodontal phase 1 therapy consisted of scaling and root planning with ultrasonic and hand instruments under local anesthesia.
  bisphosphonate therapy: bisphosphonate therapy refers to the use of zoledronic acid 5 mg/year (i.v.)
  GCF: gingival crevicular fluid collection by the same investigator.
- Group B: scaling and root planning, no bisphosphonate therapy
  periodontal phase 1 therapy: periodontal phase 1 therapy consisted of scaling and root planning with ultrasonic and hand instruments under local anesthesia.
  GCF: gingival crevicular fluid collection by the same investigator.
- Group C: bisphosphonate therapy (zoledronic acid)
  bisphosphonate therapy: bisphosphonate therapy refers to the use of zoledronic acid 5 mg/year (i.v.)
  GCF: gingival crevicular fluid collection by the same investigator.
- Group D: Systemically and periodontally healthy controls No intervention has been made
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 12 | 10 | 11 | 10
ng/ml | 1389.177 (670.834) | 1085.405 (618.136) | 1596.585 (841.026) | 2131.87 (485.78)
Statistical Analysis 1: Comparison: Group A vs Group B vs Group C vs Group D; Test type: Other; p < 0.01, Kruskal-Wallis; Mean Difference (Final Values) = 0.01

2. Primary Outcome: Dkk-1 Values for 6th Month
Description: levels of dickkopf-related protein-1 in 6th month
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Group A: * Subjects with chronic periodontitis and osteoporosis.
  * Phase 1 periodontal therapy and bisphosphonate therapy ( Aclasta: intravenous infusion of 5 mg of zoledronic acid once a year) were administered to the subjects.
  Phase 1 periodontal therapy: Scaling and root planning with ultrasonic and hand instruments under local anesthesia.
  Bisphosphonate therapy: Using aclasta: intravenous infusion of 5 mg of zoledronic acid once a year
- Group B: * Subjects with chronic periodontitis and systemically healthy.
  * Phase 1 periodontal theraphy was administered to the subjects.
  Phase 1 periodontal therapy: Scaling and root planning with ultrasonic and hand instruments under local anesthesia.
- Group C: * Subjects with periodontally healthy and osteoporosis.
  * Bisphosphonate therapy ( Aclasta: intravenous infusion of 5 mg of zoledronic acid once a year) were administered to the subjects.
  Bisphosphonate therapy: Using aclasta: intravenous infusion of 5 mg of zoledronic acid once a year
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 12 | 10 | 11 | 10
ng/ml | 3358.265 (1477.199) | 1963.185 (966.451) | 3263.665 (2298.590) | 4269.39 (1734.73)
Statistical Analysis 1: Comparison: Group A vs Group B vs Group C vs Group D; Test type: Other; p < 0.05, Kruskal-Wallis

3. Secondary Outcome: Sost Values for 12th Month
Description: levels of sclerostin in 12th month
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 12 | 10 | 11 | 10
ng/ml | 1702.265 (1012.124) | 1347.330 (876.383) | 1114.988 (368.840) | 2131.87 (485.78)
Statistical Analysis 1: Comparison: Group A vs Group B vs Group C vs Group D; Test type: Other; p < 0.05, Kruskal-Wallis

4. Secondary Outcome: Dkk-1 Values for 12th Month
Description: levels of dickkopf-related protein-1 in 12th month
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Group A: -Subjects with chronic periodontitis and osteoporosis.
- Group B: -Subjects with chronic periodontitis and systemically healthy.
- Group C: -Subjects with periodontally healthy and osteoporosis.
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 12 | 10 | 11 | 10
ng/ml | 3440.67 (2347.112) | 3203.802 (1706.081) | 2490.553 (841.512) | 4269.39 (1734.73)
Statistical Analysis 1: Comparison: Group A vs Group B vs Group C vs Group D; Test type: Other; p < 0.05, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored/assessed
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed in any participants.
Groups:
- Group A: Participants received periodontal phase 1 treatment and used bisphosphonate.
- Group B: Participants received periodontal phase 1 treatment.
- Group C: Participants used bisphosphonate.
- Group D: Participants did not receive any treatment.
Arm/Group | Group A | Group B | Group C | Group D
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT04149405/ICF_002.pdf
  • Study Protocol and Statistical Analysis Plan (2018-12-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT04149405/Prot_SAP_003.pdf